CLINICAL TRIAL: NCT00337545
Title: Phase II Trial of RAD001 in Patients With Refractory Colorectal Cancer
Brief Title: Phase II Trial of RAD001 in Refractory Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD0012467; Swedish Cancer Institute 05128
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Colorectal Cancer
Keywords: Metastatic; Refractory
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Everolimus

INTERVENTIONS:
Drug: RAD001

SUMMARY:
Single center open-label study of an oral agent (RAD001) in subjects with metastatic colorectal cancer refractory to at least 2 standard chemo/biologic regimens.

DETAILED DESCRIPTION:
Study is completed and closed.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer refractory to at least 2 chemo/biologic regimens
* Measurable disease
* ECOG 0-2

Exclusion Criteria:

* CNS disease
* Chemotherapy or radiotherapy < 4 weeks prior
* Active bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-05; Study Completion 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gold, M.D., Principal Investigator — Swedish Cancer Institute
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States